CLINICAL TRIAL: NCT02755350
Title: Demonstrating Effective Delivery of Daily Oral HIV Pre-Exposure Prophylaxis as Part of HIV Combination Prevention Intervention Among Young Women at High HIV Risk, Female Sex Workers and Men Who Have Sex With Men in Kenya (IPCP-KENYA)
Brief Title: Introducing PrEP Into HIV Combination Prevention - Kenya
Acronym: IPCP-Kenya
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LVCT Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Sex Workers Outreach Project (Unknown); National AIDS Control Council (Unknown); National AIDS and STI Control Programme (Unknown); Health Options for Young Men with AIDS/STI (Unknown); Bar Hostess Empowerment & Support Programme (Unknown); Gay and Lesbian Coalition Kenya (Other); ISHTAR MSM (Unknown); Kenya Sex Workers Alliance (Unknown); London School of Hygiene and Tropical Medicine (Other); Imperial College London (Other); Results for Development (Unknown); O' Neill Institute (Unknown); AVAC (Unknown); Nyanza Western Kenya LGBTI Coalition (Unknown); World Health Organization (Other); International AIDS Vaccine Initiative (Network); Centres for Disease Control and Prevention, Kenya. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NON-SSC NO. 456; OPP1104919 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2015-11-12; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: PrEP; HIV Prevention; combination prevention; demonstration project
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Pre-Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Truvada (Experimental): Daily oral PrEP (Truvada) is provided to a cohort of 2100 participants who will be followed up at multiple intervals, in months 1, 4, 7, 10 and 12) for 12 months. The PrEP users will attend 7 visits at the project sites over the project period. In between some visits, they will return to the pharmacy for a refill of PrEP, counselling on adherence and medication of side effects.
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Daily oral PrEP will be provided to a cohort of 2100 participants (female sex workers, men who have sex with men and young women at high HIV risk) in Kenya. Baseline data will be collected from all participants at enrolment. PrEP users will be followed up at multiple intervals, in months 1, 4, 7, 10 and 12) for 12 months. The PrEP users will attend 7 visits at the project sites over the project period and in between these visits, they will return to the pharmacy for PrEP refill, adherence counselling and assessment of side effects.
  Other Names: Pre Exposure Prophylaxis (PrEP)

SUMMARY:
Daily oral PrEP will be delivered to men who have sex with men (MSM), female sex workers (FSWs) and young women (YW) as part of a defined package of HIV combination prevention intervention for 12 months in 5 sites in Kenya. The project will assess adherence, adverse events, side effects, user satisfaction, cost, facility preparedness and provider competencies. PrEP eligibility and screening tools for MSM, YW and FSWs will be piloted and validated. Pregnant women will be enrolled in a sub-group and followed through 12 months post- partum to measure mother and infant outcomes that include health status, birth outcomes, birth defects, risk behavior and PrEP adverse effects. With lessons from initial PrEP studies in West and Central Africa, this project will apply good participatory practice guidelines through 1) continuous engagement with communities of FSWs, YW and MSM and 2) development and use of a communication engagement and advocacy strategy that will provide correct information, address attitudes and concerns whilst increasing demand for PrEP uptake. The actual cost of delivering HIV combination prevention which includes PrEP will also be assessed and cost effectiveness modeled.

DETAILED DESCRIPTION:
The project will be undertaken in 3 counties of Kenya (Nairobi, Kisumu and Homa Bay) that have high HIV prevalence. 5 sites (2 government and 3 non-governmental) have been purposively selected for the demonstration because they serve high risk populations, have existing HIV prevention services and have adequate cohort of HIV negative clients who are potential candidates for PrEP. The sites include LVCT Health's Nairobi CBD and Tivoli sites, SWOP City clinic, Homa Bay County Referral Hospital and Korogocho Health Centre. The demonstration project will use a prospective cohort design employing mixed-methods. A cohort of 2100 PrEP users (female sex workers aged 18 and above, men who have sex with men aged 18 and above, young women at high HIV risk aged 15 -29) will be followed over 12 months to assess biological and behavioral outcomes through laboratory and survey assessments. This will be complemented by review of routine service delivery statistics (to assess PrEP uptake), cost data, and qualitative data to be obtained from in-depth interviews and focus groups with health providers, PrEP users, and peer educators/community health workers at multiple points in time.This project will be implemented in a 'real life' or 'real world' setting where there will be no control or comparison arms. However, pregnant women at enrolment and female participants who become pregnant during project implementation, who choose to continue on PrEP will be enrolled in a sub-group and followed through 12 months post-partum.

Activities to be undertaken prior and during project implementation:

* HIV prevention packages, provider training, quality management and service delivery guidelines and standard operating guidelines will be developed.
* PrEP eligibility and screening tools for target populations will be piloted and validated prior to project implementation. For young women, a test of understanding will be additionally administered to screen for eligibility.
* Community sensitization and demand creation activities will be conducted prior to and during implementation. Existing peer educators for FSW and MSM from each site will reach out to these populations through hot spots. For young women at high HIV risk, outreach activities will be done by peer educators and community health volunteers (CHVs) through 1) community-based organizations which work with young women (such as youth groups, organised social gatherings [chamas], [government administrative meetings such as chief barazas] 2) political leaders such as women representatives 3) existing services reaching sexually active young women such as family planning, maternal-child health (MCH) 4) community radio and 5) anywhere that young women gather such as water points.
* To ensure adherence to good participatory practice guidelines (GPP) that outline community engagement in clinical and research activities, a national community advisory board (CAB) and community advisory committees (CAC) at each project site will be formed. The CAB and CACs will participate in the development and execution of demand creation activities, development of community education materials, peer education and mobilization, strategy development, project design, implementation and advocacy.

Project procedures:

At the screening visit, eligible and willing participants will be provided with full information about PrEP, results of efficacy trials, known side effects and potential adverse events, and daily dosing schedule. They will receive counselling on adherence to PrEP including discussions between PrEP users and service providers on developing new routines and cues as a way to facilitate good adherence. They will also receive detailed information about the project, including the number and sequence of project visits, procedures at each visit, use of MEMS Caps, and the option to discontinue PrEP use during the course of the project. They will also be counselled on available combination prevention strategies such as condom use and provided with free condoms. Participants will also be informed that PrEP will only be available for 12 months.

Willing participants will sign an informed consent form, and complete a survey questionnaire to provide baseline information on their demographics, sexual risk behaviours, risk perceptions, medical history, alcohol and drug use, contraceptive use, fertility intentions, and use of other combination HIV prevention services. They will receive HIV testing and counselling (HTC), tests for Hepatitis B surface antigen, STI syndromic screening and management as well as testing for gonorrhoea, blood draw for creatinine level and pregnancy test where applicable. Individuals who test HIV positive are ineligible for the project and will be referred to care and treatment according to standard practice. Pregnant women and women who become pregnant during the project implementation will be enrolled in a pregnancy sub group, upon their consent. Those who decline participation will receive referrals to prenatal care.

Participants will return to the project site after 14 days (2 weeks), for an enrolment visit where they will receive a one month PrEP prescription, a HIV re-test and counselling on adherence, side effects, and available supportive interventions. Participants will be asked to return after 2 weeks for assessment of adherence and side effects. They will then return to the site for the first follow up visit (1 month after enrollment visit) where they will receive the following services: counselling on HIV risk behaviours, adherence, side effects/experience with PrEP, HTC, pregnancy test (for women), creatinine level test, STI syndromic screening and management, gonorrhoea test, drug level testing, and PrEP prescription for one month (with refills from pharmacy at months 2 and 3). Every 10th participant will complete a quantitative survey at exit.

Participants will then return to the site for a quarterly visit at months 4, 7, and 10 after enrolment. The services provided during these visit will be similar to those at the first follow up visit. Participants who display high adherence will be provided with a 3 months' supply of PrEP. Those who need close monitoring will be provided with a one month's supply and will return for pharmacy refills monthly.

Participants will finally return for an exit visit, 12 months after enrolment. They will receive services similar to those at enrolment. They will also complete an exit survey, and discuss post project PrEP access with the health provider.

Individuals who want to discontinue PrEP use will be allowed to do so, and asked to consent for in depth interview to discuss their experience and decision to stop. Those who display poor adherence will be discontinued from PrEP. Those who sero-convert will be referred to care and treatment services as per standard practice.

Key strategies for retention will include 1) follow up of participants by peer educators and community health volunteers, 2) using text messages for appointment reminders and adherence support 3) enrolling participants in support groups, and 4) adherence buddies.

Indepth interviews with PrEP users and health providers, focus group discussions with peer educators, CHWs, and support group members will be conducted at Months 1, 6 and 12. The actual cost of implementing HIV combination prevention that includes PrEP will be collected throughout the project implementation period.

Ethical considerations observed in the implementation of this project include protocol approval by KEMRI ethics research committee, informed consent for participants, confidentiality of participants and their data and ensuring safety of participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported interest in and willingness to take PrEP
* Score cut-off on PrEP screening tool
* HIV- negative test at time of enrollment (per testing algorithm)
* No clinical symptoms of acute HIV infection including fever, lymphadenopathy, pharyngitis, skin rash, myalgias/arthralgias.
* Hepatitis-B virus antigen negative (upon screening)
* Creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula) (upon screening)
* Not breastfeeding
* Not currently taking PrEP or enrolled in another PrEP demonstration project
* Willingness to visit the project site of choice for follow up visits throughout the project period
* Knowledge of spoken English or Kiswahili
* Is in good general health and does not report a medical condition which may make their participation unsafe.
* Is not currently taking post exposure prophylaxis (PEP).
* Willing to provide contact information and be contacted by project staff between visits for follow up and support.
* Able to summarise the purpose of the demonstration project and their role as participants.
* Sexually active - having had sex in the last 3 months

Specific eligibility criteria for each project population are as follows:

* MSM: Age 18 and above; Self-reported anal sex with a man
* FSW: Age 18 and above; Self-identification as a sex worker;
* Young Women: Aged 15-29 ;Among young women aged 15-17, a test of understanding will also be administered to further determine their eligibility.

Exclusion Criteria:

* HIV positive
* Breastfeeding
* HIV positive
* Women above 29 years
* Those who fail test of understanding
* Those who do not meet the score cut-off on PrEP screening tool
* Not sexually active

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of young women, female sex workers and men who have sex with men correctly identified as being at high risk of HIV, in need of and willing to take PrEP. | 4 months
  Validation of tools for risk identification and indication for PrEP initiation
Proportion of men who have sex with men, female sex workers and young women at high risk of HIV enrolled into a HIV combination prevention intervention package that includes PrEP. | 4 months
  Validation of tools for risk identification and indication for PrEP initiation
Number of participants adhering to oral PrEP as measured using the MEMS cap and MedAmigo system. | 12 months
Proportion of participants enrolled and retained in a HIV combination prevention package that includes PrEP over a period of 12 months. | 12 months
Number of enrolled participants reporting side effects as recorded on the clinical and adverse event forms | 12 months
Unit cost analysis of identifying and enrolling clients on PrEP in a 'real world' setting identified through mathematical modelling | 12 months
Cost estimates for providing PrEP to high risk populations determined through cost models | 12 months
Number of enrolled participants reporting pregnancy complications as recorded on the pregnancy outcome forms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Serah N Njenga, BA, Principal Investigator — LVCT Health; Lawrence J Gelmon, MD.MPH, Principal Investigator — Sex Workers Outreach Project; Nduku S Kilonzo, PhD, Principal Investigator — National AIDS Control Council, Kenya; Helgar K Musyoki, MPH, Principal Investigator — National AIDS and STIs Control Program, Kenya
Locations (1):
- LVCT Health, Nairobi, Nairobi County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided